CLINICAL TRIAL: NCT02821013
Title: A Randomized Phase III Trial of the Duration of Anti-PD-1 Therapy in Metastatic Melanoma
Brief Title: Duration of Anti-PD-1 Therapy in Metastatic Melanoma
Acronym: STOP-GAP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Melanoma and Skin Cancer Trials Limited (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ME13; UQ-QMP-0001 (Other: QMP)
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Unresectable/Metastatic Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Intermittent PD-1 Inhibitor therapy (Active Comparator): Any PD-1 inhibitor that is commercially available, government approved and publicly funded. Dose as recommended by the manufacturer.
  Interventions: Drug: Intermittent PD-1 inhibitor therapy
- Arm 2: Continuous PD-1 Inhibitor therapy (Active Comparator): Any PD-1 inhibitor that is commercially available, government approved and publicly funded. Dose as recommended by the manufacturer.
  Interventions: Drug: Continuous PD-1 inhibitor therapy

INTERVENTIONS:
Drug: Intermittent PD-1 inhibitor therapy
  Arms: Arm 1: Intermittent PD-1 Inhibitor therapy
Drug: Continuous PD-1 inhibitor therapy
  Arms: Arm 2: Continuous PD-1 Inhibitor therapy

SUMMARY:
The purpose of this study is to compare the effects on patients with metastatic melanoma of taking a government approved and paid-for PD-1 inhibitor intermittently, with taking the same type of agent continuously. Researchers want to see if the two ways of giving this type of treatment work equally well in extending the life of patients with melanoma, or not.

DETAILED DESCRIPTION:
The standard or usual treatment for this disease is to receive treatment with a class of agents known as PD-1 inhibitors, or also with the names anti-PD-1 therapy, immunotherapy and checkpoint inhibitors. PD-1 inhibitors turn on the immune system, so that it can fight the cancer cells in the body. Clinical trials have shown that PD-1 inhibitors (such as pembrolizumab and nivolumab) can shrink tumours and extend the life of patients with melanoma.

To-date, PD-1 inhibitors have been given to patients with melanoma continuously (non-stop), for as long as they remain beneficial, for up to a total duration of 2 years. The 2 year duration was chosen because doctors thought it was reasonable, and has been adopted as the standard or usual duration because it was shown to work in clinical trials. However, some recent observations suggest that PD-1 inhibitors may work just as well if they are given for a shorter time and/or in an intermittent schedule. Intermittent means to take breaks from receiving the drug when, and for as long as, the melanoma is better.

The investigators doing this study are interested to find out whether patients with melanoma live as long when the PD-1 inhibitors are given continuously (non-stop) or in an intermittent schedule (taking breaks). If the two ways of giving the treatment were to be shown to be just as good, benefits of an intermittent schedule may include less clinic visits and side effects, better quality of life, and less cost over time for the Health Care System. However, this is not known at present.

ELIGIBILITY:
Minimum age 18 or as specified in the Product Monograph and eligible for public funding.

Inclusion Criteria:

* Histologically confirmed melanoma that is unresectable / metastatic (stage III or stage IV).
* Eligible to receive treatment with a government approved and publically-funded PD-1 inhibitor, according to the guidance / indications described in the Product Monograph / Provincial Formulary.
* Patients must have evidence of unresectable / metastatic disease, that is considered evaluable by the investigator and can be followed, but measurable disease is not mandatory.
* Patients with brain metastases are allowed, provided they are stable according to the following definitions:

  1. Without evidence of progression for at least four weeks prior to randomization and have no evidence of new or enlarging brain metastases.
  2. Treated with surgery and without evidence of progression prior to randomization and have no evidence of new or enlarging brain metastases.
  3. Treated with stereotactic radiosurgery and without evidence of progression prior to randomization and have no evidence of new or enlarging brain metastases.
* Patient is able (i.e. sufficiently fluent) and willing to complete the quality of life and health utility questionnaires in either English or French. The baseline assessment must be completed within required timelines, prior to randomization. Inability (lack of comprehension in English or French, or other equivalent reason such as cognitive issues or lack of competency) to complete the questionnaires will not make the patient ineligible for the study. However, ability but unwillingness to complete the questionnaires will make the patient ineligible.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate.
* Patients must be accessible for treatment and follow-up. Investigators must assure themselves the patients randomized on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.
* Patients must be randomized prior to the start of, or within 16 weeks from, the initiation of PD-1 inhibitor treatment. For patients who are being randomized before the start of treatment, the PD-1 inhibitor should be started within 5 working days after randomization. Patients who initiate treatment with combination anti-PD-1 and anti-CTLA-4 therapies who experience toxicity may be randomized at the time prior to starting single-agent PD-1 inhibitor. Repeat imaging must be done within 50 days prior to randomization to ensure the patient has no evidence of disease progression

Exclusion Criteria:

* Patients not willing to stop anti-PD-1 therapy, if randomized to the intermittent arm.
* Patients with any contraindications to PD-1 inhibitors, as described in the Product Monograph or Provincial Formulary, and/or not eligible to receive anti-PD-1 therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Estimated)
Dates: Start 2016-10-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 7 years

SECONDARY OUTCOMES:
Progression-free survival using RECIST 1.1 / Immune-Related RECIST (irRECIST) | 7 years
Response rate using RECIST 1.1 / Immune-Related RECIST (irRECIST) | 7 years
Duration of response using RECIST 1.1 / Immune-Related RECIST (irRECIST) | 7 years
Number and severity of adverse events using CTCAE v 4.0 | 7 years
Quality of Life measured by EORTC QLQ-C30 | 7 years
Economic evaluation consisting of both healthcare utilization and health utilities measured by the EQ-5D questionnaire | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Xinni Song, Study Chair — Ottawa Hospital Research Institute; Tara Baetz, Study Chair — Cancer Centre of Southeastern Ontario at Kingston
Locations (31):
- Australia (12):
  - Mildura Base Public Hospital, Victoria, Mildura
  - Coffs Habour Health Campus - NCCI, Coffs Harbour, New South Wales
  - Riverina Cancer Care Centre Wagga Wagga, Wagga Wagga, New South Wales
  - Calvary Mater Newcastle Hospital, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Cairns Hospital, Cairns, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - The Queen Elizabeth Hospital, Woodville, South A.
  - Monash Medical Centre, Clayton, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Royal Brisbane and Womens Hospital, Herston
- Canada (19):
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Surrey, Surrey, British Columbia
  - BCCA - Vancouver, Vancouver, British Columbia
  - BCCA - Victoria, Victoria, British Columbia
  - Horizon Health Network, Fredericton, New Brunswick
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Health Sciences North, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Waterloo Regional Health Network (WRHN), Kitchener, Ontario
  - London Health Sciences Centre Research Inc., London, Ontario
  - Trillium Health Partners - Credit Valley Hospital, Mississauga, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - The Research Institute of the McGill University, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No